CLINICAL TRIAL: NCT02234336
Title: Assessment of Wall Thickness in Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Patricia A. Pellikka, Professor of Medicine, College of Medicine, Mayo Clinic
Other Study IDs: 14-004757
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Echocardiography; hypertrophic cardiomyopathy; cardiomyopathy; magnetic resonance imaging; contrast
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with HCM: All subjects will undergo noncontrast echocardiography, contrast echocardiography and cardiac MRI.
  Interventions: Procedure: Noncontrast echocardiography; Procedure: Contrast Echocardiography; Procedure: Cardiac magnetic resonance imaging

INTERVENTIONS:
Procedure: Noncontrast echocardiography
Procedure: Contrast Echocardiography
Procedure: Cardiac magnetic resonance imaging

SUMMARY:
Assessment of wall thickness in hypertrophic cardiomyopathy (HCM) is of diagnostic and prognostic importance given its known association with sudden cardiac death. However, data regarding comparison of imaging modalities for this key measurement is lacking. This study seeks to compare assessment of maximum wall thickness between clinically indicated echocardiography (with and without contrast) and clinically indicated cardiac magnetic resonance imaging.

DETAILED DESCRIPTION:
Patients receiving clinically indicated echocardiograms and cardiac magnetic resonance imaging at Mayo Clinic will be eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically and echocardiographically defined hypertrophic cardiomyopathy.
2. Clinically indicated transthoracic echocardiography as part of the medical evaluation.
3. No contradiction to administration of ultrasonic echocardiography contrast.
4. Planned clinically indicated cardiac magnetic resonance imaging as part of medical evaluation.
5. No contraindication to cardiac magnetic resonance imaging (such as cochlear implants, central nervous system aneurysm clips and other implanted medical devices).
6. Age 18 years and older

Exclusion Criteria:

1) Insufficient image quality for determination of maximal wall thickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hypertrophic cardiomyopathy (HCM)
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Wall Thickness | approximately 1 week after enrollment
  All subjects will undergo noncontrast echocardiography, contrast echocardiography and cardiac MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pellikka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States